CLINICAL TRIAL: NCT07168551
Title: Association of Hyperuricemia and Non Alcoholic Fatty Liver Disease and Liver Fibrosis Risk in Adult Obese Patients
Brief Title: Is There a Relationship Between Uric Acid Level and Liver Fibrosis in Obese Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Adel Mahmoud Abu Shady, Internal medicine Resident doctor, Assiut University
Other Study IDs: UNLF
Record Dates: First submitted 2025-08-27; First posted 2025-09-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Hyperuricemia; NAFLD (Nonalcoholic Fatty Liver Disease); Liver Fibrosis
MeSH Terms: conditions — Hyperuricemia; Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — Hematologic Tests; Liver Function Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1- obese +-nafld+- fibrosis: Obese patients with non alcoholic fatty liver disease with fibrosis
  Interventions: Diagnostic Test: *Lab Methods:* 1- Serum Uric Acid levels 2-Liver Function Tests 3- Lipid Profile . 4- Haemoglobin A1c level . 5- Serum glucose level .; Radiation: *Imaging Studies:* 1- Ultrasound 2 - FibroScan; Device: Instruments:* 1- *Automated Analyzers*: Used for blood tests, such as serum uric acid and liver function tests.
- obese +- hyperuricemia +- nfld+- fibrosis: Obese patients with hyperuricemia and non alcoholic liver disease and fibrosis
  Interventions: Diagnostic Test: *Lab Methods:* 1- Serum Uric Acid levels 2-Liver Function Tests 3- Lipid Profile . 4- Haemoglobin A1c level . 5- Serum glucose level .; Radiation: *Imaging Studies:* 1- Ultrasound 2 - FibroScan; Device: Instruments:* 1- *Automated Analyzers*: Used for blood tests, such as serum uric acid and liver function tests.
- Healthy controls: Healthy controls
  Interventions: Diagnostic Test: *Lab Methods:* 1- Serum Uric Acid levels 2-Liver Function Tests 3- Lipid Profile . 4- Haemoglobin A1c level . 5- Serum glucose level .; Radiation: *Imaging Studies:* 1- Ultrasound 2 - FibroScan; Device: Instruments:* 1- *Automated Analyzers*: Used for blood tests, such as serum uric acid and liver function tests.

INTERVENTIONS:
Diagnostic Test: *Lab Methods:* 1- Serum Uric Acid levels 2-Liver Function Tests 3- Lipid Profile . 4- Haemoglobin A1c level . 5- Serum glucose level . — Lab methods
Radiation: *Imaging Studies:* 1- Ultrasound 2 - FibroScan — Imaging
Device: Instruments:* 1- *Automated Analyzers*: Used for blood tests, such as serum uric acid and liver function tests. — Instrument

SUMMARY:
1. Identifying the association between hyperuricemia and NAFLD can lead to early detection and prevention of liver fibrosis in adult obese patients.
2. Understanding the relationship between hyperuricemia and NAFLD can inform targeted therapy, such as urate-lowering treatment, to potentially slow disease progression.

3 - To examine the relationship between serum uric acid levels and liver fibrosis severity*: Assessing the correlation between serum uric acid levels and the severity of liver fibrosis in adult obese patients with NAFLD.

4- To identify potential mechanisms underlying the association*: Exploring the potential mechanisms by which hyperuricemia may contribute to the development and progression of NAFLD and liver fibrosis in adult obese patients.

DETAILED DESCRIPTION:
Hyperuricemia is associated with nonalcoholic fatty liver disease (NAFLD), whereas whether the association differed by hyperuricemia onset age remained unclear. This study sought to investigate the associations of hyperuricemia onset age with the risk of incident NAFLD across adulthood.

Obesity has been demonstrated to show a consistent link with the increased possibility of nonalcoholic fatty liver disease (NAFLD). Since both serum uric acid (SUA) and obesity are essential components of metabolic syndrome (MetS), it is uncertain whether the incidence of NAFLD results from serum uric acid, obesity, or other potential factors based on previous studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Adults (typically 18-65 years old)

2 - Body Mass Index (BMI): Obese patients with a BMI ≥ 30 kg/m²

3- Hyperuricemia : Elevated serum uric acid levels (typically > 7 mg/dL for men and > 6 mg/dL for women)

Exclusion Criteria:

* excessive alcohol consumption ( > 20 gm /day in men and 10 in g /day in women )

  2- use of steatogenic within the past 6 months

  3- positive test for hepatitis B surface antigen and hepatitis B core antibody

  4- Drug induced liver injury and autoimmune hepatitis

  5 - cirrhosis and other causes of liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult obese patients
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NAFLD | 1 year
  The proportion of adult obese patients with NAFLD in the study population

SECONDARY OUTCOMES:
Serum uric acid level | 1 year
  The serum uric acid level in adult obese patients